CLINICAL TRIAL: NCT06604091
Title: Cohort Profile：The Shandong Adenomyosis Cohort of Population Undergoing Reproductive Technology (SAart)
Status: Active, not recruiting | Type: Observational
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Linlin Cui, Professor, The Second Hospital of Shandong University
Other Study IDs: KYLL2024742
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Adenomyosis; in Vitro Fertilization
Keywords: adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Mild adenomyosis group: disease extent :< 25% of uterine volume affected by adenomyosis
  Interventions: Other: Treatment protocol
- Moderate adenomyosis group: disease extent: 25-50% of uterine volume affected by adenomyosis
  Interventions: Other: Treatment protocol
- Severe adenomyosis group: disease extent: > 50% of uterine volume affected by adenomyosis
  Interventions: Other: Treatment protocol
- Control group: Receiving IVF treatment because of common factor, such as fallopian tube factors
  Interventions: Other: Treatment protocol

INTERVENTIONS:
Other: Treatment protocol — Treatment options for ovarian stimulation include long-acting and antagonist regimens and other ovulation induction regimens. Options for frozen embryo transfer include natural protocols, mild ovarian stimulation regimens, hormone replacement therapy (HRT) regimens, and down-regulated combined HRT regimens. The treatment regimen is refined in the above protocol. The treatment of patients follows the principles of real-world clinical practice.

SUMMARY:
Previous studies have shown that compared with infertile women without adenomyosis, the clinical pregnancy rate, live birth rate and continuous pregnancy rate of women with adenomyosis significantly reduce, and the abortion rate obviously increased. However, these studies lack a definite classification of adenomyosis, so the true effect of adenomyosis with different severity on pregnancy outcomes are not clear. Our research team intends to collect clinical data of infertility patients with adenomyosis receiving IVF and the detailed classification of adenomyosis according to MUSA criteria. Finally, we can have an objective recognition of adenomyosis on pregnancy outcomes, which also bring benefits to evidence-based clinical practice.

DETAILED DESCRIPTION:
Previous studies have shown that compared with infertile women without adenomyosis, the clinical pregnancy rate, live birth rate and continuous pregnancy rate of women with adenomyosis significantly reduce, and the abortion rate obviously increased. However, these studies lack a definite classification of adenomyosis, so the true effect of adenomyosis with different severity on pregnancy outcomes are not clear. Our research team intends to collect clinical data of infertility patients with adenomyosis receiving IVF and the detailed classification of adenomyosis according to MUSA and ultrasound consensus. Finally, we can have an objective recognition of adenomyosis on pregnancy outcomes, which also bring benefits to evidence-based clinical practice.

The detailed inclusion and exclusion criteria are as follows:

Inclusion criteria

1.Age of all participants ≥ 20 and < 38 years. 2.Receiving IVF treatment because of adenomyosis or other common factor, such as fallopian tube factors.

3.Conforming to MUSA criteria. 4. Body mass index < 30 kg/m2. 5.The level of AMH ≥ 0.8 ng/ml. Exclusion criteria

1. Uterine fibroids (International Federation of Gynecology and Obstetrics (FIGO) type 0--I--II or type III--IV fibroids > 3 cm).
2. Untreated endometrial polyps, hydrosalpinx or uterine adhesions.
3. RSA or RIF.
4. Intracytoplasmic sperm injection (ICSI) and preimplantation genetic testing (PGT).
5. Concurrent and/or recent involvement in other research within previous 3 months of study enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Age of all participants ≥ 20 and< 38 years.
2. Receiving IVF treatment because of adenomyosis or other common factor, such as fallopian tube factors.
3. Conforming to MUSA criteria.
4. Body mass index < 30 kg/m2.
5. The level of AMH ≥ 0.8 ng/ml.

Exclusion Criteria:

1. Uterine fibroids (International Federation of Gynecology and Obstetrics (FIGO) type 0--I--II or type III--IV fibroids < 3 cm).
2. Untreated endometrial polyps, hydrosalpinges or uterine adhesions.
3. RSA or RIF.
4. Intracytoplasmic sperm injection (ICSI) and preimplantation genetic testing (PGT).
5. Concurrent and/or recent involvement in other research within previous 3 months of study

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This trial aims to evaluate the impact of uterine adenomyosis on the pregnancy outcomes of patients undergoing IVF for assisted conception. The study population consists of individuals aged 20-38 years, diagnosed with uterine adenomyosis or general assisted conception patients, diagnosed by ultrasound to meet the MUSA criteria, with a BMI of less than 30 kg/m2, an AMH level of ≥ 0.8 ng/ml, excluding those with uterine fibroids, untreated intrauterine space-occupying lesions, and diseases such as RSA and RIF, and who have not received ICSI and PGT treatments.
Sampling Method: Non-Probability Sample
Enrollment: 2241 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
cumulative live birth rate | from pregnancy to delivery
  The numerator is number of live births from fresh or frozen embryo transfer in one ovarian stimulation cycle. More than one live birth is considered as one live birth. Denominator is defined as patients who have undergone oocyte retrieval and have either achieved at least one live birth or who have no surplus embryos.

SECONDARY OUTCOMES:
implantation rate | from transplantation to delivery
  IR is the ratio of the total number of gestational sacs confirmed by TVUS to the total number of transferred embryos.
biochemical pregnancy rate | from transplantation to pregnancy
  Serum β-hCG level ≥ 10 mIU/mL is defined as biochemical pregnancy.
ectopic pregnancy rate | from transplantation to clinical pregnancy
  Ectopic pregnancy is defined as the presence of extra-uterine gestational sacs or masses.
miscarriage rate | pregnancy loss before 28 gestational weeks
  Miscarriages mean pregnancy loss before 28 gestational weeks. Clinical pregnancy loss ≤ 12 gestational weeks is an early miscarriage, and pregnancy loss between 12 and 28 gestational weeks is a late miscarriage.
clinical pregnancy rate | pregnancy loss before 28 gestational weeks
  Clinical pregnancy is defined as visible intra-uterine pregnancy or extra-uterine pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Lin l Cui, M.D., Ph.D., Study Chair — The Second Hospital of Shandong University, China
Locations (1):
- The Second Clinical Hospital of Shandong University, Jinan, Shandong, China